CLINICAL TRIAL: NCT04405947
Title: Randomized Prospective Study Comparing Reversed Shoulder Prosthesis Through the Superior Anterior Approach and the Deltopectoral Approach
Brief Title: Influenze of Approach in Reversed Shoulder Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Carlos Torrens, Principal investigator, Hospital del Mar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/7913/I
Record Dates: First submitted 2020-05-20; First posted 2020-05-28 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Outcomes Assessments, Patients; Rotator Cuff Arthropathy
Keywords: reverse shoulder arthroplasty; scapular notch; deltopectoral; anterosuperior approach

STUDY DESIGN:
Intervention Model Description: prospective randomized study
Who Masked: Outcomes Assessor
Masking Description: given the fact that the different approaches come with different scars, just the outcomes assessor can be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- deltopectoral (Other): deltopectoral surgical approach
  Interventions: Procedure: Reverse Shoulder Arthroplasty
- antero-superior (Other): antero-superior approach
  Interventions: Procedure: Reverse Shoulder Arthroplasty

INTERVENTIONS:
Procedure: Reverse Shoulder Arthroplasty — implantation of a reversed shoulder prostheses through two different surgical approaches

SUMMARY:
To determine the differences in the placement of the glenoid implant of the inverted prostheses when they are implanted using a superior approach and using an anterior approach.

DETAILED DESCRIPTION:
Inverted prostheses have proven to be effective in the treatment of all those pathologies that involve a deterioration of the rotator cuff (secondary arthropathy, acute fractures, sequelae of fractures, tumor surgery and revision surgery). Despite this, numerous complications have been described after the use of inverted prostheses, such as glenoid erosion, infections, dislocation, or aseptic loosening. The most frequent complication related to the use of inverted prostheses is glenoid erosion that can occur in up to 96% of cases. This complication appears early in the evolution, usually before 2 years after surgery. Its clinical significance is not yet clear, but it seems that it may be a cause of long-term prosthetic loosening. To avoid the development of glenoid erosion, the best option is to place the glenoid component low, so that if the glenoid component is flush with the lower margin of the glena, the chances of developing glenoid erosion are significantly reduced. Two types of approaches have been used to implant these prostheses, the deltopectoral and the superior anterior approach. Each of them has its advantages and disadvantages, so that deltopectoral seems to improve surgical exposure and therefore favors the best placement of the glenoid component, but sacrifices the subscapularis tendon, increasing the risk of dislocation of the components. On the contrary, the superior anterior approach respects the subscapularis tendon, reducing the risk of dislocation of the components but gives worse surgical exposure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with secondary osteoarthritis of the shoulder who are candidates for an inverted prosthesis
* Acute fractures <2 weeks of evolution in patients candidates for inverted prostheses
* No previous surgeries of the affected shoulder
* Acceptance by the patient to participate in the study

Exclusion Criteria:

* Fractures> 2 weeks of evolution
* Previous surgeries on the affected shoulder
* Not signing the informed consent
* Cognitive impairment
* Institutionalization of the patient

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-01-13 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2020-10-29 (Actual)

PRIMARY OUTCOMES:
positioning of the metaglene of the reverse shoulder prostheses | 2 years
  to determine the metaglene postioning in both surgical approaches by measuring the distance between the inferior part of the metaglene and the glenoid inferior rim. The measurement will be done in an AP X-ray view of the shoulder and with the help of the measure tool in the PACS system of viewing.

SECONDARY OUTCOMES:
scapular notch | 2 years
  determine scapular notch development in both approaches as determined with the aid of an AP X-ray view of the shoulder and thus classifying the scapular notch development according to Sirveaux et al. classification system.
functional outcome | 2 years. The minimum value of the Constant Score is 0 and the maximum is 100. The higher scores mean a better outcome.
  determine the functional outcome as measured with the Constant Score at 2-years follow-up